CLINICAL TRIAL: NCT03537768
Title: A Multi-center, Randomized Study of the Efficacy of Ulipristal Acetate (UPA) 30 mg, Levonorgestrel (LNG) 1.5 mg, and LNG 3.0 mg for Emergency Contraception (EC) in Women With Weight ≥ 80 kg
Brief Title: Study Comparing Emergency Contraception Effectiveness in Women Who Weight ≥ 80 kg
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We weren't seeing as many pregnancies we initially thought.
Sponsor: Kimberly Myer (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Kimberly Myer, Program Director, Premier Research
Organization: Premier Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCN013C
Record Dates: First submitted 2018-04-17; First posted 2018-05-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-08

CONDITIONS: Contraception
MeSH Terms: interventions — ulipristal acetate; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- UPA 30mg (Active Comparator)
  Interventions: Drug: Ulipristal Acetate
- LNG 1.5 mg (Active Comparator)
  Interventions: Drug: Levonorgestrel
- LNG 3.0 (Active Comparator)
  Interventions: Drug: Levonorgestrel

INTERVENTIONS:
Drug: Ulipristal Acetate — UPA Tablet
  Other Names: Ella
  Arms: UPA 30mg
Drug: Levonorgestrel — LNG Tablet
  Other Names: Plan B
  Arms: LNG 1.5 mg
Drug: Levonorgestrel — LNG Tablet (x2)
  Other Names: Plan B (double dose)
  Arms: LNG 3.0

SUMMARY:
The proposed research study is a Phase IIb, multi-center, single-blind, randomized study of UPA 30 mg, LNG 1.5 mg and LNG 3.0 mg to evaluate EC effectiveness in women with weight ≥ 80 kg who present within 72 hours of unprotected intercourse.

DETAILED DESCRIPTION:
Orally-dosed emergency contraception (EC) is highly effective when used properly. EC is up to 90% effective at preventing pregnancy following unprotected intercourse. Both ulipristal acetate (UPA) and levonorgestrel (LNG) delay or inhibit ovulation when used for EC. For individual women, use of EC provides a critical backup to prevent unintended pregnancy.

However, obesity may severely impair EC effectiveness. Data from two large randomized control trials to identify risk factors for EC failure. A woman of obese body mass index (BMI) (≥30mg/kg2) using LNG-based EC had more than a 4 times greater risk of pregnancy compared to her normal BMI counterpart and a woman of overweight BMI (25-29.9) was at twice the risk of pregnancy. Failure was also associated with a high body weight. LNG-based EC appears to have a ceiling of efficacy at 70 kg and no efficacy for women 80 kg and above. It is believed that by doubling the dose to LNG 3.0 mg, serum levels of LNG are corrected to a therapeutic range.

ELIGIBILITY:
Inclusion Criteria:

1. Be in good general overall health with no chronic medical conditions that result in periodic exacerbations that require significant medical care.
2. Between 18 and 40 years inclusive at the enrollment visit.
3. Weight ≥ 80 kg.
4. Have regular menstrual cycles that typically occur every 21-35 days when not using hormonal contraception.
5. If subject is postpartum or post-abortal, she must have experienced a menstrual bleed since the pregnancy ended
6. If a subject recently used non-injectable hormonal contraception, one bleeding episode consistent with menses must have occurred since last use;
7. Willing to avoid use of any hormonal or intrauterine contraception until the end of the study;
8. For women with a recent history of Depo Provera use, the most recent injection must have been at least 6 months before study entry, and the subject must have had at least one normal menstrual cycle (2 consecutive menses);
9. Request emergency contraception within 72 hours (3 days) after unprotected coitus, as defined by lack of contraceptive use, condom breakage (including condoms lubricated with spermicide), or other barrier contraceptive method failure;
10. Have a negative urine pregnancy test at time of screening
11. Reports all acts of unprotected coitus since her prior menses are within 72 hours prior to enrollment;
12. Willing to abstain from further acts of unprotected intercourse until the end of the study;
13. Give voluntary, written informed consent, and agree to observe all study requirements including being available for follow up for at least the next 4 weeks;
14. Accepts that the risk of pregnancy with oral EC is greater than that following placement of a copper IUD for EC.

Exclusion Criteria:

1. Be currently pregnant (positive high-sensitivity urine pregnancy test);
2. Be currently breastfeeding or within 30 days of discontinuing breastfeeding, unless the subject has already had a menses following discontinuation of breastfeeding;
3. Desire to use hormonal systemic contraception within 5 days of study drug use
4. Have had a female sterilization procedure;
5. Have a partner with a history of vasectomy;
6. Current inability to tolerate oral medication;
7. Have impaired hypothalamic-pituitary-adrenal reserve or oral glucocorticoid replacement therapy in the last year.
8. Have known liver disease;
9. Have known liver abnormalities with elevated enzymes at least twice the upper limit of normal requiring use of liver enzyme inducers.
10. Have known hypersensitivity to the active substance UPA or LNG, or any of the excipients of the study treatment.
11. Have a current need for exogenous hormones.
12. Have concomitant use of strong CYP3A4 inhibitors (as identified by the FDA) or inducers at the time of or planned use within 3 days of dosing;
13. Use any medications that can interfere with the metabolism of hormonal contraceptives; take antibiotics that can interfere with metabolism of hormonal contraceptives at the time of or planned use within 3 days of dosing of the study drug; or use any drugs designated by the FDA as falling in the Pregnancy and Lactation narrative subsections (formerly Category D or X medications).
14. Current or recent (within one month) participation in any other trial of an investigational medicine or device or planning to participate in another clinical trial during this study.
15. Have a history of a bariatric surgery procedure associated with malabsorption.
16. Live outside of the catchment area of the study site.
17. Have used UPA or LNG EC within 30 days prior to enrollment and not had a menses since using the drug.
18. Be a site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities. -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 532 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of pregnancies of UPA 30 mg, LNG 1.5 mg and LNG 3.0 mg in women with weight ≥ 80 kg for emergency contraception (within 72 hours of unprotected intercourse). | 1-3 months

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events of UPA 30 mg, LNG 1.5 mg and LNG 3.0 mg in women with weight ≥80 kg seeking emergency contraception. | 1-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Diana Blithe, PhD, Study Director — NICHD Director
Locations (18):
- United States (18):
  - Essential Access Health, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Hawaii, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Bellevue Hospital Center, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati-Holmes Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland MacDonald Women's Hospital, Cleveland, Ohio
  - Oregon Health Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh/Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelman A, Jensen JT, Brown J, Thomas M, Archer DF, Schreiber CA, Teal S, Westhoff C, Dart C, Blithe DL. Emergency contraception for individuals weighing 80 kg or greater: A randomized trial of 30 mg ulipristal acetate and 1.5 mg or 3.0 mg levonorgestrel. Contraception. 2024 Sep;137:110474. doi: 10.1016/j.contraception.2024.110474. Epub 2024 Apr 23. PMID 38663539